CLINICAL TRIAL: NCT06153641
Title: Cytokeratin 18 a Novel Non-invasive Biomarker for Rejection in Liver Transplant Patients
Brief Title: Cytokeratin 18 Non-invasive Biomarker for Rejection in Liver Transplant Patients
Status: Active, not recruiting | Type: Observational
Sponsor: St. Louis University (Other)
Collaborators: Mid-America Transplant (Other)
Responsible Party: Principal Investigator, Ajay Jain MD, Division Director of Pediatric Gastroenterology and Hepatology, St. Louis University
Other Study IDs: 29508
Record Dates: First submitted 2023-11-20; First posted 2023-12-01 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Liver Transplant Rejection; Liver Transplant Failure and Rejection
Keywords: Liver Transplant; Stable post liver transplant; Post transplant liver biopsy; Healthy nontransplant without liver disease
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum collected from 5ml of blood will be stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Biopsy arm: Post-transplant patients undergoing standard of care liver biopsy (Biopsy arm).
  Interventions: Other: N/A-Observational Study
- Stable post-liver transplant arm: Stable post-liver transplantation patients without rejection (Stable post-liver transplant arm).
  Interventions: Other: N/A-Observational Study
- Healthy arm: Healthy non-transplant control patients without liver disease (Healthy arm).
  Interventions: Other: N/A-Observational Study

INTERVENTIONS:
Other: N/A-Observational Study — N/A-Observational Study

SUMMARY:
Liver transplantation is a lifesaving procedure; however, there are chances that the body may reject the organ following liver transplantation, and this remains a significant concern. This rejection of the transplanted, healthy liver tissue further adds to the patient's illness and also increases the related costs of treatment. Currently, liver biopsy is the standard procedure used for diagnosing this rejection. Being an invasive procedure (requiring the introduction of instruments into the body), this procedure also increases the chances of death of the patient. Researchers are looking into the identification of testing methods that can act as a sign of this rejection without requiring the introduction of instruments into the body. This type of testing could also allow for adjusting the doses of drugs given to the patient to decrease the chances of graft failure.

A particular event that occurs during rejection in the body is the death of liver cells. Thus, tracking cell death using a blood test would be an important tool in assessing rejection. CK-18 is a protein in the liver cells that is thought to be linked to the changes occurring as a result of cell death. This study will be looking into a new idea of measuring CK-18 levels and compare them to an existing index to develop a reliable test for liver transplant rejection without introducing any instruments into the body.

The purpose of this research study is to assess the history and collect blood samples to be tested for measuring CK-18 levels and assess certain other markers in the blood.

DETAILED DESCRIPTION:
Cellular rejection following liver transplantation is of worldwide occurrence and a major cause of morbidity affecting 15 to 20 percent of liver transplantation recipients. Elevation of serum aminotransferase may be suspicious of rejection and typically precedes clinical symptoms of fever and jaundice. However, such clinical signs as well biochemical parameters are neither specific nor sensitive for detection of rejection or its degree of severity.

The current standard of care remains a liver biopsy for confirmation of transplant rejection. While significant procedural advances have been made, liver biopsy is an invasive procedure, requiring sedation, and has a small but definite risk of complications including mortality. Developing noninvasive biomarkers which could mitigate the need for an invasive liver biopsy remains a major national and international research focus in the field of hepatology. This could also lay the foundation for early non-invasive longitudinal tracking of rejection and help in decreasing graft failure.

Cytokeratin 18 is a cytoskeletal protein found in hepatocytes and is thought to be a major intermediate filament protein linked to the morphological changes of cell death. During hepatocyte apoptosis, cytokeratin 18 is cleaved by caspases. The resulting novel neo-epitope occurs specifically during apoptosis and represents apoptotic cell death. M30 a monoclonal antibody recognizes this cleaved epitope (CK-18) and thus serves as a novel biomarker for apoptosis. Apoptosis is a known event in rejection. Several mechanisms have been postulated to lead to apoptosis during rejection which include granule-exocytosis pathway, the Fas-mediated pathway and induction by cytokines. Additionally, there appears to be a significant co-relation between the grade of rejection and severity of apoptosis.

These observations lead us into the exciting possibility that CK-18 measurements could prove to be a very valuable noninvasive biomarker for hepatic cellular rejection and could pave the path towards predictive models tracking rejection and its progression. The purpose of this research study is to collect blood samples to be tested for measuring CK-18 levels, assess certain other markers in the blood, and assess the history.

Approximately 105 patients will be enrolled in this study at Saint Louis University.

This is a prospective study that includes three specific cohorts of subjects as follows (no randomization of subjects):

1. Post-transplant patients undergoing standard-of-care liver biopsy (Biopsy arm).
2. Stable post-liver transplantation patients without rejection (Stable post-liver transplant arm).
3. Healthy non-transplant control patients without liver disease (Healthy arm).

Each participant will be assigned a unique participant ID at the time of enrollment. All participants' data and samples collected will be saved by this unique participant ID. All blood samples will be labeled with a study number and sent for assessment of CK-18 levels and other markers to understand rejection.

A participant may spend less than one hour on this research study (the time it takes to give consent, review medical information, and have their blood drawn).

Reviewing their medical records will collect Information about participants (age, race, gender) and their health. The research team will try to take the research blood sample when participants already have a blood test done for their regular health checks, but there may be times when the participant must have blood drawn just for the study.

The blood sample required for this research study will be collected as follows, depending on the participant category may fall into:

1. If the participant is a healthy patient or a participant who underwent liver transplantation and is stable post-transplantation with no symptoms and signs of rejection. In that case, the research sample will be collected with the standard of care lab work they will have as a part of routine healthcare. If such is not possible, the Participant may need to get an extra stick.
2. If a participant is undergoing a liver biopsy. In that case, an intravenous line is usually placed as a standard of care at participating centers at the time of liver biopsy - especially in the pediatric population. Research blood would be collected during line placement or with standard-of-care lab work.

If such cannot be obtained, then the research-only blood sample would be collected. There may be times when the research team is unable to get adequate blood for our research study at this time, which is when participants may need to have additional blood drawn for the study.

Participants may be re-enrolled in the study more than once if they qualify. Participants will be asked if they are willing to participate each time and will be re-consented each time.

* If a participant has a liver transplant after completing participation in the healthy arm, the Participant may be eligible for re-enrollment in the study under other arms (Stable post-liver transplant arm or biopsy arm).
* If a participant has an episode of rejection and is scheduled for liver biopsy after completing participation in the stable post-liver transplant arm, the participant may be eligible for re-enrollment in the study under the biopsy arm since this study captures the rejection events.
* If a participant has a subsequent episode of rejection and is scheduled for another liver biopsy after completing participation in the biopsy arm, the Participant may be eligible for re-enrollment in the study under the liver biopsy arm since this study captures the rejection events.
* If a participant get stable in the study doctor's opinion after completing participation in the biopsy arm. The participant may be eligible for re-enrollment in the study under the stable post-liver transplant arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be at least 1 year of age at enrollment.
* There shall be no restrictions regarding sex, race or ethnicity
* All Patients who have received a liver transplant will be approached for enrollment in the study.

Study Group-Specific Inclusion Criteria:

• The patients who are scheduled for a liver biopsy for suspicion of liver transplant rejection (Biopsy arm).

Note-1: If a patient gets a subsequent episode of rejection and the patient is scheduled for another liver biopsy after completing participation in the biopsy arm, it will make the patient eligible for re-enrollment in the study under the biopsy arm since this study captures the rejection events. The patient will be re-consented each time and given a new participant ID each time.

Note-2: If the patient gets stable in the study doctor's opinion after completing participation in the biopsy arm, it will make the patient eligible for re-enrollment in the study under the stable post-liver transplant arm. The patient will be re-consented and given a new participant ID.

Control Group specific inclusion Criteria:

• Healthy non transplant controls(Healthy arm).

Note-1: If a patient gets a liver transplant after completing participation in a healthy arm, it will make the patient eligible for re-enrollment in the study under other arms (stable post-liver transplant arm or biopsy arm). The patient will be re-consented each time and given a new participant ID each time.

• Liver transplant recipients without rejection: Patients who are 'stable' post liver transplantation would be approached (Stable post-liver transplant arm).

Note-1: If a patient gets an episode of rejection after completing participation in the stable arm, it will make the patient eligible for re-enrollment in the study under the biopsy arm since this study captures the rejection events. The patient will be re-consented each time and given a new participant ID each time.

Exclusion Criteria for All Arms:

1. Known infectious hepatitis
2. Patient non-compliant
3. For patients with any unforeseen risk factors, all efforts will be made to not enroll them in the study. If a patient has exceeded the 50mL/3mL per kg limit clinically, the patient will not be enrolled in the study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Three specific cohorts of subjects as follows (no randomization of subjects):
  1. Post-transplant patients undergoing standard of care liver biopsy (Biopsy arm).
  2. Stable post-liver transplantation patients without rejection (Stable post-liver transplant arm).
  3. Healthy non-transplant control patients without liver disease (Healthy arm).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Characterize baseline CK-18 levels in healthy non transplant control patients and 'stable' post transplantation patients without rejection. | through study completion, an average of 1 year
  Characterize baseline CK-18 levels in healthy non transplant control patients and 'stable' post transplantation patients without rejection.
Determine cross-sectional relationship between CK-18 levels and severity of rejection. | through study completion, an average of 1 year
  Determine cross-sectional relationship between CK-18 levels and severity of rejection.
Ultimate goal would be to determine if serial CK-18 assessment could longitudinally predict rejection and its progression. | through study completion, an average of 1 year
  Our ultimate goal would be to determine if serial CK-18 assessment could longitudinally

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Jain, MD, Principal Investigator — Saint Louis University/SSM Health Cardinal Glennon Children's Hospital
Locations (1):
- SSM Health Cardinal Glennon Children's Hospital & Saint Louis University Hospital (SSM Health- SLU Hospital), St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided